CLINICAL TRIAL: NCT04995978
Title: Insulin Resistance in Men With Prostate Cancer on Androgen Deprivation Therapy
Brief Title: Insulin Resistance and Androgen Deprivation Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were recruited and the study was deemed not feasible
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Sandeep Singh Dhindsa, M.D., F.A.C.E, Professor of Medicine, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 31991
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Prostate Cancer; Insulin Resistance
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: Pioglitazone 30 mg
- placebo (Placebo Comparator)
  Interventions: Drug: placebo tablet

INTERVENTIONS:
Drug: Pioglitazone 30 mg — Subjects will self-administer a 30 mg pioglitazone oral tablet daily for 6 months.
  For patient taking a diabetic regimen of gemfibrozil, the dose will be 15 mg daily.
  Arms: Pioglitazone
Drug: placebo tablet — Subjects will self-administer an oral placebo tablet containing cellulose daily for 6 months.
  Arms: placebo

SUMMARY:
Prostate cancer is the most common malignancy amongst men in United States. Androgen deprivation therapy (ADT) with long acting gonadotropin releasing hormone agonists is routinely used as adjuvant therapy in intermediate and high risk localized or locally advanced prostate cancer. Since ADT induces insulin resistance and diabetes, it is important that cellular and molecular effects of ADT are investigated to define precisely the mechanisms involved in the pathogenesis of insulin resistance. Pioglitazone, a known insulin sensitizer, may provide amelioration of insulin resistance in these patients.

DETAILED DESCRIPTION:
Investigators plan to conduct a prospective, randomized, double-blind, placebo-controlled trial in 44 men with nonmetastatic prostate cancer who are receiving ADT with long acting GnRH agonist (study group). Study subjects will undergo insulin clamp, subcutaneous fat biopsy, muscle biopsy, have a blood sample taken and fibroscan performed prior to randomization of study drug. They will then be randomized to 30 mg pioglitazone or placebo tablet daily for 6 months. Blood samples will be drawn 2 and 4 months following the initiation of the study drug. The final study visit will be at 6 months. Subjects will undergo clamp, fat biopsy, muscle biopsy, blood sampling, fibroscan and will be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer, non-metastatic
* Have been on ADT with long acting GnRH agonist continuously for last 3 months, AND planning to continue ADT for at least 6 months

Exclusion Criteria:

* Used pioglitazone in last 6 months
* Heart Failure NYHA Class 3 or 4
* Known to have osteoporosis at this time.
* history of bladder cancer
* Hemoglobin <8 g/dl
* eGFR <15 ml/min/1.73m2
* liver enzymes (ALT or AST) >3 times the upper limit of normal

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | 6 months
  The primary endpoint of the study is to detect a difference in insulin sensitivity as measured by whole body glucose uptake during clamps after treatment with pioglitazone as compared to placebo.

SECONDARY OUTCOMES:
Insulin signaling (Insulin receptor substrate expression in fat tissue) | 6 months
  A secondary endpoint for the study will be comparison of the relative change from baseline in insulin signaling after pioglitazone or placebo.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis Univeristy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No